CLINICAL TRIAL: NCT03273348
Title: Role of Oncoplastic Breast Surgery In Breast Cancer Treatement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alaa Mohammed Sebaiy, general surgery specialist, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17200114
Record Dates: First submitted 2017-08-25; First posted 2017-09-06 (Actual); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammaplasty

STUDY DESIGN:
Intervention Model Description: This study aim to evaluate the outcome on oncological side and patient satisfaction on the aesthetic side with skin-sparing mastectomy and immediate breast reconstruction for patients with early breast cancer .
  .
  The obtained results may contribute to the formulation of guidelines achieving low morbidity, high levels of patient satisfaction and oncological safety in breast cancer patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- oncoplastic breast surgery (Other): This study aim to evaluate the outcome on oncological side and patient satisfaction on the aesthetic side with skin-sparing mastectomy and immediate breast reconstruction for patients with early breast cancer .
  Interventions: Procedure: Oncoplastic breast surgery

INTERVENTIONS:
Procedure: Oncoplastic breast surgery — , Skin sparing mastectomy and immediate breast reconstruction will be conducted to all women included in the study, transverse rectus abdominis musculocutaneous flap recostruction and latissimus dorsi myocutaneous pedicle-flap with and without implant
  Other Names: breast reconstruction

SUMMARY:
Role of Oncoplastic Breast Surgery In Breast Cancer Treatement

DETAILED DESCRIPTION:
Breast cancer is the most common cancer in women throughout the world (FerlayJ.,2010) .

The overarching principle guiding surgical management of women with breast cancer remains the oncological safety. The mainstay of satisfactory local control continues to be adequate clearance of the primary tumour and involved axillary lymph nodes. Improvements in understanding of tumour biology have enabled the risk of loco-regional recurrence and distant events to be further reduced by adjuvant, or neo-adjuvant, radiotherapy and systemic treatments. In keeping with this, breast conserving therapy has become well established as the treatment of choice for most women with early breast cancer . However, approximately one-third of women still undergo mastectomy, either due to patient preference or in cases where breast conservation is not oncologically or aesthetically compatible with the size or distribution of disease. (Reefy et al; 2010)

The primary aim of BCS is preservation of the breast while adhering to oncologic principles, with the secondary objective to provide breast aesthetics. In recent years, with advances in early detection and adjuvant therapy life expectancy has prolonged in breast cancer prolonged and quality of life issues have gained importance (Veiga DF.,2010)

Skin sparing mastectomy involves the en-bloc removal of all glandular tissue including the nipple-areola complex and in some cases adjacent biopsy scars and skin overlying superficial tumours. In contrast to conventional mastectomy, there is maximal preservation of the remaining breast skin envelope and infra-mammary fold that facilitate immediate breast reconstruction with autologous tissue and/or prosthetic implants by utilising the native skin envelope to optimise the contour, texture, colour and scarring of the reconstructed breast. (Cunnick and Mokbel; 2004).

Due to the positive results obtained in the surgical treatment of breast cancer, the prevalence of this technique is increasing throughout the world and our country. There was an approximately 2.3-fold increase in OBS publications over the last five years (Losken A et al.,2014)

Surgical planning and timing of reconstruction should include breast volume, tumor location, the extent of glandular tissue resected, enabling each patient to receive an individual "custom-made" reconstruction. With immediate oncoplastic approach, the surgical process is smooth since oncological and reconstructive surgery can be associated in one operative setting. Additionally, because there is no scar and fibrosis tissue, breast reshaping is easier, and the aesthetic is improved (Munhoz AM et al .,2011) When considering a patient for an oncoplastic breast conserving procedure, the following points must be considered:

1. volume of tissue to be excised;
2. tumour location;
3. breast size and glandular density;
4. patient related risk factors, particularly smoking, obesity, diabetes, previous surgery;
5. adjuvant therapies. Excision volume is the single, most predictive factor for breast deformity (Clough KB et al .,2010).

Recently, several studies have contributed to the evidence base supporting the oncological adequacy of skin sparing mastectomy in selected early-stage breast cancer , excluding inflammatory breast cancer and tumours with extensive involvement of the skin. In this study the oncological safety, post-operative morbidity and patients' satisfaction with skin sparing mastectomy and immediate breast reconstruction will be evaluated in a prospective cohort of women with early-stage breast cancer. (Cunnick and Mokbel; 2004) Skin sparing mastectomy and immediate breast reconstruction is particularly attractive for women with ductal Carcinoma In-Situ in view of the fact that post-mastectomy radiotherapy is not given to the reconstructed breast and the risk of loco-regional recurrence is very low. (Spiegel and Butler; 2003)

Most women who will undergo skin sparing mastectomy and immediate breast reconstruction for early-stage breast cancer will not require post-mastectomy radiotherapy. However, post-mastectomy radiotherapy has been shown to reduce loco-regional recurrence and improve survival for patients with three or more involved regional lymph nodes or tumors >5 cm. (Recht and Edge; 2003) Mastectomy can also be indicated in several non-invasive conditions. Ductal Carcinoma In-Situ may necessitate mastectomy when the lesions are extensive, multi-centric or recurrent, however, patients request to be managed in this way. Mastectomy for ductal Carcinoma In-Situ is associated with cure rates in excess of 98%. (Mokbel; 2003)

ELIGIBILITY:
Inclusion Criteria:

* The study will include 30 women with early-stage breast cancer treated at general surgery department, Assuit University Hospitals
* For all patients an informed consent for their inclusion in the study including the use of images will be obtained.
* Selection criteria include women with a pre-operative diagnosis (clinical examination, imaging and needle biopsy) of Tis, T1 and T2 tumours without extensive skin involvement.

Exclusion Criteria:

* • contraindaction for general anesthesia

  * Positive margin requiring mastectomy
  * Insufficient remaining breast volume
  * Diffuse microcalcifications
  * Multicentric tumor?
  * Inflammatory breast cancer
  * Previous radiotherapy
  * Concomitant disease ( Diabetes, smoking )

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2017-09-28 (Estimated); Primary Completion 2019-09-28 (Estimated); Study Completion 2019-10-28 (Estimated)

PRIMARY OUTCOMES:
oncological safety | for 2 weaks
  the pathological report postoperative reveals safety free margins

SECONDARY OUTCOMES:
postoperative recurrence of malignany | assess for 1 year postoperative
  follow up any malignancy recurrence post operative by MRI , Mammograghy and look for any new skin nodule appearance
mortality rate | up to 3 months postoperative for each case
  number of deaths intraoperative and postoperative related to surgery
post operative skin edge ischemia | assess for 1 month postoperative
  look for any postoperative ischemia appear in the skin flap as appearance of dark unhealthy tissue in the edge

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
postoperative imaging such as mammogram, ultrasound and MRI studies

REFERENCES:
- [Background] Ferlay J, Shin HR, Bray F, Forman D, Mathers C, Parkin DM. Estimates of worldwide burden of cancer in 2008: GLOBOCAN 2008. Int J Cancer. 2010 Dec 15;127(12):2893-917. doi: 10.1002/ijc.25516. PMID 21351269
- [Background] Veiga DF, Veiga-Filho J, Ribeiro LM, Archangelo I Jr, Balbino PF, Caetano LV, Novo NF, Ferreira LM. Quality-of-life and self-esteem outcomes after oncoplastic breast-conserving surgery. Plast Reconstr Surg. 2010 Mar;125(3):811-7. doi: 10.1097/PRS.0b013e3181ccdac5. PMID 20195109 (Retraction: PMID 30880791 J Cancer Res Ther. 2019 Jan-Mar;15(1):264)
- [Background] Losken A, Dugal CS, Styblo TM, Carlson GW. A meta-analysis comparing breast conservation therapy alone to the oncoplastic technique. Ann Plast Surg. 2014 Feb;72(2):145-9. doi: 10.1097/SAP.0b013e3182605598. PMID 23503430